CLINICAL TRIAL: NCT01420926
Title: A Randomized Phase II Trial of Decitabine-Based Induction Strategies for Patients >/= 60 Years Old With Acute Myeloid Leukemia (AML)
Brief Title: Decitabine With or Without Bortezomib in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02987; NCI-2011-02987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000709218; CALGB-11002 (Other: Alliance for Clinical Trials in Oncology); CALGB-11002 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Bortezomib; Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (decitabine) (Experimental): REMISSION INDUCTION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-10. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR CRi proceed to continuation therapy. Patients achieving CR or CRi proceed to maintenance therapy.
  CONTINUATION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (decitabine and bortezomib) (Experimental): REMISSION INDUCTION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 2-11 and 1.3 mg/m^2 bortezomib SC on days 1, 4, 8, and 11. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR or CRi proceed to continuation therapy. Patients achieving CR or CRi proceed to maintenance therapy.
  CONTINUATION THERAPY: Patients receive 1.3 mg/m^2 bortezomib SC on day 1 and 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive 1.3 mg/m^2 bortezomib SC on day 1 and 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm B (decitabine and bortezomib)
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well giving decitabine with or without bortezomib works in treating older patients with acute myeloid leukemia. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells,by stopping them from dividing, or by stopping them from spreading. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether decitabine works better when given with or without bortezomib in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if treatment of older acute myeloid leukemia (AML) patients with decitabine and bortezomib significantly improves the overall survival times of older AML patients compared with decitabine alone.

SECONDARY OBJECTIVES:

I. To determine the rate of complete remission (CR and CR + incomplete blood count recovery [CRi]) for each of the 2 treatment regimens in the proposal.

II. To determine the overall survival, progression-free survival, disease-free survival and for each of the treatment regimens on this study.

III. To determine whether ongoing treatment with these regimens prolongs overall survival even in the absence of complete remission.

IV. To describe the frequency and severity of adverse events, as well as the tolerability of each of these regimens in patients treated on this study.

V. To describe the interaction of pretreatment disease and patient characteristics including morphology, cytogenetics, molecular genetics, white blood cell (WBC) count, blood and bone marrow blast count, age, performance status and comprehensive geriatric assessment on clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: REMISSION INDUCTION THERAPY: Patients receive decitabine intravenously (IV) over 1 hour once daily (QD) on days 1-10. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR or CR with CRi proceed to continuation therapy. Patients achieving CR or CR with CRi proceed to maintenance therapy.

CONTINUATION THERAPY: Patients receive decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: REMISSION INDUCTION THERAPY: Patients receive decitabine IV over 1 hour QD on days 2-11 and bortezomib subcutaneously (SC) on days 1, 4, 8, and 11. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR or CRi proceed to continuation therapy. Patients achieving CR or CR with CRi proceed to maintenance therapy.

CONTINUATION THERAPY: Patients receive bortezomib SC on day 1 and decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive bortezomib SC on day 1 and decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 2 years, every 3 months for 2 years, and then once a year for a maximum of 10 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal pathologic diagnosis of AML (>= 20% blasts in the bone marrow based on World Health Organization [WHO] criteria) EXCLUDING:

  * Acute promyelocytic leukemia t(15;17)(q22;q12); PML-RARA
  * Acute myeloid leukemia with t(8;21)(q22;q22); RUNX1-RUNXT1 as determined by the Ohio State University (OSU) Molecular Reference Laboratory, per Cancer and Leukemia Group B (CALGB) 20202; however patients who (1) are >= 75 years; and/or (2) have an ejection fraction of < 40%; and/or (3) have a performance status of > 2, may be registered to CALGB 20202 and registered and treated on CALGB 11002 prior to receiving the FLT3 mutation and core-binding factor (CBF) molecular screening results from CALGB 20202
  * Acute myeloid leukemia with inv(16)(p13.1;q22) or t(16;16)(p13.1;q22); CBFB-MYH11 as determined by the OSU Molecular Reference Laboratory, per CALGB 20202; however patients who (1) are >= 75 years; and/or (2) have an ejection fraction of < 40%; and/or (3) have a performance status of > 2, may be registered to CALGB 20202 and registered and treated on CALGB 11002 prior to receiving the FLT3 mutation and CBF molecular screening results from CALGB 20202
* Absence of FLT3 mutation (ITD or point mutation) determined by the OSU Molecular Reference Laboratory, per CALGB 20202; however patients who (1) are >= 75 years; and/or (2) have an ejection fraction of < 40%; and/or (3) have a performance status of > 2, may be registered to CALGB 20202 and registered and treated on CALGB 11002 prior to receiving the FLT3 mutation and CBF molecular screening results from CALGB 20202
* No prior treatment for AML except:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea
  * Cranial radiotherapy (RT) for central nervous system (CNS) leukostasis (one dose only)
  * Growth factor/cytokine support
* AML patients with an antecedent hematologic disorder (AHD) or myelodysplastic syndrome (MDS) are eligible for this trial provided that they have not received treatment for their AHD or MDS with cytotoxic chemotherapy (e.g., cytarabine, daunorubicin, etc.), decitabine, or bortezomib; patients may have been previously treated with azacitidine if their last dose was >= 90 days prior to starting 11002
* AML patients with therapy-related myeloid neoplasms (t-MN) are eligible if they have not received radiation therapy or chemotherapy (not including hormonal therapy) for their primary malignancy or disorder for > 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail J Roboz, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (53):
- United States (53):
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Hartford Hospital, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Ritchie EK, Klepin HD, Storrick E, Major B, Le-Rademacher J, Wadleigh M, Walker A, Larson RA, Roboz GJ. Geriatric assessment for older adults receiving less-intensive therapy for acute myeloid leukemia: report of CALGB 361101. Blood Adv. 2022 Jun 28;6(12):3812-3820. doi: 10.1182/bloodadvances.2021006872. PMID 35420672
- [Derived] Roboz GJ, Mandrekar SJ, Desai P, Laumann K, Walker AR, Wang ES, Kolitz JE, Powell BL, Attar EC, Stock W, Bloomfield CD, Kohlschmidt J, Mrozek K, Hassane DC, Garraway L, Jane-Valbuena J, Baltay M, Tracy A, Marcucci G, Stone RM, Larson RA. Randomized trial of 10 days of decitabine +/- bortezomib in untreated older patients with AML: CALGB 11002 (Alliance). Blood Adv. 2018 Dec 26;2(24):3608-3617. doi: 10.1182/bloodadvances.2018023689. PMID 30567725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 165 participants were enrolled from 24 sites from November 2011 to March 2013
Pre-assignment Details: Two (2) participants never received any protocol treatment; per study design these patients were excluded from all analyses.
Groups:
- Arm I (Decitabine): REMISSION INDUCTION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-10. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR or CRi proceed to continuation therapy. Patients achieving CR or CRi proceed to maintenance therapy.
  CONTINUATION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Decitabine and Bortezomib): REMISSION INDUCTION THERAPY: Patients receive 20 mg/m^2 decitabine IV over 1 hour QD on days 2-11 and 1.3 mg/m^2 bortezomib SC on days 1, 4, 8, and 11. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving CR or CRi proceed to continuation therapy. Patients achieving CR or CRi proceed to maintenance therapy.
  CONTINUATION THERAPY: Patients receive 1.3 mg/m^2 bortezomib SC on day 1 and 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive 1.3 mg/m^2 bortezomib SC on day 1 and 20 mg/m^2 decitabine IV over 1 hour QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Started | 82 | 81
Completed | 22 | 18
Not Completed | 60 | 63
Not completed — Adverse Event | 6 | 4
Not completed — Death | 18 | 17
Not completed — Withdrawal by Subject | 11 | 17
Not completed — Non-protocol treatment | 17 | 20
Not completed — Physician Decision | 8 | 5

BASELINE CHARACTERISTICS:
Population: Two (2) participants never received any protocol treatment; per study design these patients were excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib) | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Median (Full Range); unit: years] | 72.4 [60.7 to 92.3] | 72.9 [60.5 to 90] | 72.4 [60.5 to 92.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 19 | 50
  Male | 51 | 62 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 77 | 77 | 154
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 4 | 7
  White | 74 | 73 | 147
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 163

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: Overall survival (OS) was defined as the time from study entry to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Number analyzed (Participants) | 82 | 81
months | 9.3 [5.8 to 12.2] | 8.8 [3.8 to 14.3]
Statistical Analysis 1: Comparison: Arm I (Decitabine) vs Arm II (Decitabine and Bortezomib); Test type: Superiority or Other; p = 0.30, Stratified 1-sided log-rank

2. Secondary Outcome: Complete Remission Rate (CR and CRi)
Description: Defined as the number of patients who achieve a CR or CRi divided by the total number of evaluable patients. A Complete remission (CR) requires: <5% marrow blast, > 200 nucleated cells, no blasts with auer rods, no extramedullary disease, ANC >1,000/mm^3 and platelets > 100,000/mm^3. A CR with incomplete blood count recovery (CRi) is defined as CR with exception of ANC < 1,000/mm^3 or platelets < 100,000/mm^3.
Time Frame: 48 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Number analyzed (Participants) | 82 | 81
percentage of participants | 40 [30 to 52] | 38 [28 to 50]

3. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease free survival (DFS) was defined as the time from CR to relapse or death. Relapse free and surviving patients were censored at the date of last follow-up. The median DFS with 95% CI was estimated using the Kaplan Meier method. Relapse is defined as the reappearance of blood blasts or >= 5% marrow blasts after achieving a CR or CRi.
Time Frame: 48 months
Population: Only participants who achieved a CR are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Number analyzed (Participants) | 15 | 17
months | 8.5 [3.9 to 21.3] | 15.3 [7.9 to 25.5]

4. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was defined as the time from study entry to progression or death. Progression free and surviving patients were censored at the date of last follow-up. The median DFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Number analyzed (Participants) | 82 | 81
months | 7.3 [5.3 to 8.9] | 8.0 [3.8 to 12.2]

5. Secondary Outcome: Adverse Events
Description: Adverse Events: Incidence of adverse events, assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Adverse events were collected every cycle during treatment and up to one month after treatment. Adverse events were summarized using summary statistics and frequency tables for each separate cohort. Per protocol, analysis was descriptive in nature. In this section, the number of patients that reported a grade 4 or higher event are summarized. A complete listing of Adverse Events is provided in the Adverse Events section below.
Time Frame: 48 months
Population: The 4 participants were not evaluated for adverse events were excluded from this analysis.
Measure: Number; unit: participants
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
Number analyzed (Participants) | 80 | 79
participants | 51 | 45

ADVERSE EVENTS:
Time Frame: 48 months
Description: 159 participants were evaluable for adverse events.
Arm/Group | Arm I (Decitabine) | Arm II (Decitabine and Bortezomib)
All-Cause Mortality (participants affected / at risk) | 70/82 | 75/83
Serious Adverse Events (participants affected / at risk) | 43/80 | 45/79
Other Adverse Events (participants affected / at risk) | 66/80 | 61/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Decitabine) (N=80) | Arm II (Decitabine and Bortezomib) (N=79)
Anemia (Blood and lymphatic system disorders) | 40 (51) | 39 (52)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (4) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (23) | 23 (24)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac disorders - Other (Cardiac disorders) | 3 (4) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 2 (3)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2) | 3 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 9 (12) | 7 (10)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (6) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Congenital, familial and genetic disorders - Other (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 4 (4)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (20) | 16 (19)
Diarrhea (Gastrointestinal disorders) | 14 (17) | 22 (24)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (9) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (4) | 5 (7)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 5 (5) | 2 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 21 (25) | 21 (24)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (18) | 14 (17)
Chills (General disorders) | 9 (11) | 8 (9)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 17 (19) | 23 (28)
Edema trunk (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 29 (38) | 27 (35)
Fever (General disorders) | 7 (10) | 9 (12)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 3 (3) | 3 (3)
Hypothermia (General disorders) | 0 (0) | 3 (3)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (4) | 2 (3)
Multi-organ failure (General disorders) | 3 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 6 (8)
Pain (General disorders) | 8 (8) | 8 (9)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (2) | 5 (5)
Cecal infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 8 (9) | 11 (11)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 14 (18) | 13 (16)
Mucosal infection (Infections and infestations) | 3 (5) | 2 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 12 (13) | 9 (9)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 5 (5) | 4 (4)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 6 (6) | 8 (8)
Alanine aminotransferase increased (Investigations) | 13 (15) | 15 (19)
Alkaline phosphatase increased (Investigations) | 8 (11) | 12 (14)
Aspartate aminotransferase increased (Investigations) | 15 (17) | 20 (22)
Blood bilirubin increased (Investigations) | 21 (24) | 10 (10)
Cardiac troponin I increased (Investigations) | 1 (1) | 4 (4)
Cholesterol high (Investigations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 17 (17) | 19 (26)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 6 (7) | 6 (6)
GGT increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 5 (5) | 7 (7)
Investigations - Other (Investigations) | 1 (1) | 5 (5)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 14 (18) | 17 (25)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 37 (47) | 38 (51)
Platelet count decreased (Investigations) | 39 (47) | 37 (48)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 4 (5) | 5 (6)
Weight loss (Investigations) | 7 (12) | 8 (12)
White blood cell decreased (Investigations) | 20 (27) | 18 (25)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Alkalosis (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 16 (21) | 18 (24)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (33) | 25 (33)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (7) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 (28) | 26 (32)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (21) | 19 (23)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 17 (24) | 21 (29)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (21) | 7 (8)
Hyponatremia (Metabolism and nutrition disorders) | 20 (25) | 19 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (11) | 8 (9)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 (16) | 9 (14)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (8)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (6)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (4) | 0 (0)
Dizziness (Nervous system disorders) | 9 (10) | 10 (11)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 4 (5)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 11 (12)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 3 (3)
Lethargy (Nervous system disorders) | 4 (5) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 4 (4) | 4 (4)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 9 (14)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 2 (3)
Sinus pain (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 5 (5) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Agitation (Psychiatric disorders) | 3 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (7) | 7 (7)
Confusion (Psychiatric disorders) | 7 (12) | 9 (9)
Delirium (Psychiatric disorders) | 6 (6) | 4 (4)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 6 (6) | 6 (9)
Hallucinations (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 10 (11) | 10 (11)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 7 (9) | 7 (12)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 5 (7) | 8 (8)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal calculi (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 6 (6) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 4 (5)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 13 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 23 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 12 (14)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Purpura (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (11)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 (9) | 11 (12)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (6) | 11 (12)
Hypotension (Vascular disorders) | 16 (17) | 17 (19)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 6 (6) | 3 (3)
Vascular disorders - Other (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Decitabine) (N=80) | Arm II (Decitabine and Bortezomib) (N=79)
Anemia (Blood and lymphatic system disorders) | 63 (253) | 59 (239)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3 (13) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 6 (7) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 34 (53) | 33 (45)
Leukocytosis (Blood and lymphatic system disorders) | 4 (8) | 3 (6)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 6 (7)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (3)
Cardiac disorders - Other (Cardiac disorders) | 2 (2) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 2 (3) | 3 (8)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2) | 4 (6)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 2 (3)
Pericardial effusion (Cardiac disorders) | 1 (2) | 5 (7)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 9 (11) | 6 (14)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (4)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 3 (6)
Blurred vision (Eye disorders) | 4 (24) | 6 (12)
Conjunctivitis (Eye disorders) | 2 (3) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other (Eye disorders) | 2 (5) | 4 (4)
Eye pain (Eye disorders) | 1 (1) | 1 (9)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 15 (23)
Anal pain (Gastrointestinal disorders) | 5 (6) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3) | 4 (8)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 38 (78) | 34 (65)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 34 (60) | 33 (48)
Dry mouth (Gastrointestinal disorders) | 5 (6) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 4 (8)
Dysphagia (Gastrointestinal disorders) | 7 (8) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (18) | 5 (6)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 (5) | 7 (10)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 2 (5)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 6 (7) | 7 (7)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 14 (19) | 13 (16)
Nausea (Gastrointestinal disorders) | 34 (67) | 34 (95)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 8 (11) | 4 (4)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (17) | 20 (36)
Chills (General disorders) | 9 (19) | 16 (21)
Edema face (General disorders) | 0 (0) | 4 (4)
Edema limbs (General disorders) | 32 (58) | 25 (51)
Edema trunk (General disorders) | 2 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 2 (4)
Fatigue (General disorders) | 53 (173) | 51 (170)
Fever (General disorders) | 15 (16) | 8 (10)
Flu like symptoms (General disorders) | 0 (0) | 2 (5)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 8 (9) | 8 (10)
Infusion related reaction (General disorders) | 2 (3) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (3)
Localized edema (General disorders) | 3 (3) | 2 (2)
Malaise (General disorders) | 5 (6) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (3) | 7 (8)
Pain (General disorders) | 10 (23) | 10 (14)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 3 (3)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 2 (2) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (5) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 7 (7) | 11 (14)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 14 (23) | 12 (14)
Mucosal infection (Infections and infestations) | 3 (3) | 1 (1)
Nail infection (Infections and infestations) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 1 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (2)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (4)
Sinusitis (Infections and infestations) | 5 (5) | 3 (6)
Skin infection (Infections and infestations) | 9 (11) | 10 (17)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (6) | 1 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 8 (10)
Wound infection (Infections and infestations) | 3 (5) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 12 (23) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 10 (12)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 5 (7) | 9 (17)
Alanine aminotransferase increased (Investigations) | 22 (38) | 19 (44)
Alkaline phosphatase increased (Investigations) | 17 (34) | 15 (29)
Aspartate aminotransferase increased (Investigations) | 28 (40) | 27 (54)
Blood bilirubin increased (Investigations) | 20 (44) | 12 (16)
Blood prolactin abnormal (Investigations) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 2 (2)
Cholesterol high (Investigations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 15 (26) | 20 (62)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (3) | 5 (8)
GGT increased (Investigations) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 2 (7) | 2 (2)
INR increased (Investigations) | 10 (25) | 13 (23)
Investigations - Other (Investigations) | 5 (20) | 5 (26)
Lymphocyte count decreased (Investigations) | 19 (45) | 18 (54)
Lymphocyte count increased (Investigations) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 62 (266) | 56 (224)
Platelet count decreased (Investigations) | 62 (233) | 59 (236)
Weight gain (Investigations) | 4 (7) | 3 (4)
Weight loss (Investigations) | 14 (31) | 12 (36)
White blood cell decreased (Investigations) | 30 (125) | 29 (98)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 32 (56) | 30 (78)
Dehydration (Metabolism and nutrition disorders) | 3 (6) | 4 (11)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 40 (114) | 38 (122)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 7 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 4 (7) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 33 (89) | 37 (94)
Hypocalcemia (Metabolism and nutrition disorders) | 27 (56) | 25 (66)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 5 (15)
Hypokalemia (Metabolism and nutrition disorders) | 25 (40) | 26 (46)
Hypomagnesemia (Metabolism and nutrition disorders) | 14 (33) | 13 (19)
Hyponatremia (Metabolism and nutrition disorders) | 24 (63) | 26 (48)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (16) | 11 (14)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3 (7) | 4 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (26) | 4 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (18) | 16 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 8 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 22 (39) | 14 (40)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 8 (18) | 5 (7)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 7 (24)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (18) | 9 (17)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Arachnoiditis (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (5) | 2 (3)
Dizziness (Nervous system disorders) | 13 (22) | 22 (37)
Dysgeusia (Nervous system disorders) | 3 (7) | 6 (13)
Headache (Nervous system disorders) | 15 (22) | 22 (30)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (3) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 5 (8) | 4 (9)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (8)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 19 (60)
Presyncope (Nervous system disorders) | 0 (0) | 6 (10)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 4 (7)
Tremor (Nervous system disorders) | 1 (1) | 2 (3)
Agitation (Psychiatric disorders) | 1 (1) | 1 (2)
Anxiety (Psychiatric disorders) | 9 (24) | 9 (15)
Confusion (Psychiatric disorders) | 8 (10) | 7 (8)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 13 (23) | 9 (24)
Hallucinations (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 15 (32) | 12 (23)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 6 (14) | 5 (28)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (6) | 6 (9)
Hemoglobinuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (4) | 6 (8)
Renal and urinary disorders - Other (Renal and urinary disorders) | 4 (6) | 2 (3)
Renal calculi (Renal and urinary disorders) | 1 (4) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 4 (5) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (4) | 4 (5)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 3 (4)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (45) | 16 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 (75) | 33 (63)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (10)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 10 (21) | 8 (10)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (11)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (5)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (9)
Purpura (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 25 (35) | 21 (32)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 16 (29) | 16 (25)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5)
Surgical and medical procedures - Other (Surgical and medical procedures) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 4 (5) | 2 (2)
Hypertension (Vascular disorders) | 11 (21) | 12 (17)
Hypotension (Vascular disorders) | 16 (20) | 26 (41)
Phlebitis (Vascular disorders) | 3 (3) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5) | 3 (4)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less